CLINICAL TRIAL: NCT05605093
Title: Strategies and Treatments for Respiratory Infections & Viral Emergencies (STRIVE): Shionogi Protease Inhibitor
Brief Title: Strategies and Treatments for Respiratory Infections & Viral Emergencies (STRIVE): Shionogi Protease Inhibitor (Ensitrelvir)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB closed due to futility.
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-217622
Record Dates: First submitted 2022-10-28; First posted 2022-11-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ensitrelvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- S-217622 (ensitrelvir) plus standard of care (SOC) (Experimental): Study investigational agent (ensitrelvir) will be administered as oral tablets with dosing of 375mg (3 tabs) once on Day 0 and 125mg (1 tab) once daily on Days 1-4. All participants will receive the full 5-day course, including those who are discharged from hospitalization prior to Day 4.
  Interventions: Drug: Shionogi Protease Inhibitor (S-217622)
- placebo plus standard of care (SOC) (Placebo Comparator): Study investigational placebo will be administered as oral tablets with dosing of 375mg (3 tabs) once on Day 0 and 125mg (1 tab) once daily on Days 1-4. All participants will receive the full 5-day course, including those who are discharged from hospitalization prior to Day 4.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Shionogi Protease Inhibitor (S-217622) — S-217622 (ensitrelvir) is an oral anti-SARS-CoV2 PI that does not require ritonavir co-administration The dose is 375/125 (375 mg on Day 0, followed by 125 mg daily on Days 1-4).
  Other Names: ensitrelvir
  Arms: S-217622 (ensitrelvir) plus standard of care (SOC)
Drug: placebo — Placebo is an oral tablet administered once (3 tabs) on Day 0 and once (1 tab) daily on days 1-4, 5-day course.
  Arms: placebo plus standard of care (SOC)

SUMMARY:
Treatments are needed to improve outcomes among patients hospitalized for COVID-19, including direct-acting antiviral (DAA) agents to mitigate the pathology driven by ongoing viral replication. This trial will evaluate S-217622 (ensitrelvir), an anti-SARS-CoV2 3C-like protease inhibitor (PI) developed by Shionogi &; Co. Ltd.

The study design is a randomized, placebo-controlled, multi-center international clinical trial that will evaluate the clinical efficacy of ensitrelvir when given in addition to standard of care (SOC) for inpatients with COVID-19. The SOC will be determined by local established guidelines and may include additional DAA (e.g., remdesivir) and immunomodulatory treatment strategies. Certain SOC treatments will be pre-specified prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Informed consent for trial participation.
* Hospital admission (or boarding in an emergency department or other area awaiting hospital admission) with signs and/or symptoms of a respiratory infection.
* Confirmation of SARS-CoV2 infection by nucleic acid test (NAT) or equivalent non- NAT test [list of approved tests is in the PIM] collected within the prior 14 days.
* Onset of symptoms attributable to SARS-CoV2 infection occurred within 14 days before randomization.
* Hospitalized for the management of COVID-19, with signs and/or symptoms suggestive of lower respiratory tract infection.

Exclusion Criteria:

* The patient is expected to be discharged from the hospital within the next 24 hours.
* Medical condition other than the acute respiratory infection (and its manifestations) that is likely to result in death within 7 days of randomization.
* Use of a strong CYP3A inducer within 14 days prior to enrollment
* Moribund condition, defined as prior cardiac arrest during this hospitalization and life expectancy less than 48 hours of randomization.
* Patient undergoing comfort care measures only such that treatment focuses on end-of- life symptom management over prolongation of life.
* Expected inability or unwillingness to participate in study procedures.
* In the opinion of the investigator, participation in a trial is not in the best interest of the patient.
* Allergy to investigational agent or vehicle
* Use of a concomitant medication that is contraindicated due to a drug-drug interaction with S-217622
* Moderate to severe hepatic impairment (i.e., Child-Pugh class B or C) or acute liver failure.
* Known estimated glomerular filtration rate (eGRF) <30 mL/min/1.73m 2
* Continuous renal replacement therapy or chronic dialysis
* Current pregnancy
* Current breastfeeding and unwillingness to defer breastfeeding for 30 days after the last dose of investigational agent.
* Women of child-bearing potential who are unwilling to abstain from sexual intercourse with men or practice appropriate contraception through 30 days from the last dose of the investigational agent.
* Men who are unwilling to abstain from sexual intercourse with women of child- bearing potential or to use barrier contraception through 30 days from the last dose of the investigational agent.
* Inability to take investigational agent in tablet form by mouth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Days to Recovery Scale assessed over 60 days (DRS-60) | 60 days post-intervention
  DRS-60 is a version of the STRIVE clinical recovery scale (CRS) which combines time to recovery with non-recovered clinical state and death to an ordinal outcome.0 indicates best results, 60 represents recovered on Day 60, with not recovered by Day 60 coded as 61 and death (worst outcome) as 62.

SECONDARY OUTCOMES:
mortality | 60 days post-treatment
  proportion of participants who died by Day 60
a 3-category ordinal outcome | 60 days post-treatment
  the following categories: recovered (alive and at home at Day 60), alive and not recovered, and dead
time to recovery | 60 days post-treatment
proportion of participants who died or required new invasive mechanical ventilation | 60 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cavan Reilly, PhD, Principal Investigator — University of Minnesota; Jason Baker, MD, Study Chair — University of Minnesota
Locations (187):
- United States (103):
  - University of Alabama Birmingham University Hospital (Site 213-002), Birmingham, Alabama
  - Banner University Medical Center Tucson (Site 206-004), Tucson, Arizona
  - Southern Arizona VA Healthcare System (Site 074-009), Tucson, Arizona
  - UCSF Fresno (Site 203-005), Fresno, California
  - VA Loma Linda Healthcare System (Site 074-017), Loma Linda, California
  - MemorialCare Health System (Site 066-003, Long Beach, California
  - VA Long Beach Healthcare System (Site 074-026), Long Beach, California
  - Cedars-Sinai Medical Center (Site 208-002), Los Angeles, California
  - Ronald Reagan UCLA Medical Center (Site 203-002), Los Angeles, California
  - VA Northern California Health Care System (Site 074-023), Mather, California
  - Hoag Memorial Hospital Presbyterian (Site 080-026), Newport Beach, California
  - Veterans Affairs Palo Alto Health Care System (VAPAHCS) (Site 074-005), Palo Alto, California
  - UC Davis Health (Site 203-004), Sacramento, California
  - VA San Diego Healthcare System (Site 074-016), San Diego, California
  - Zuckerberg San Francisco General Hospital and Trauma Center (Site 213-007), San Francisco, California
  - UCSF Medical Center at Mount Zion (203-007), San Francisco, California
  - San Francisco VAMC (Site 074-002), San Francisco, California
  - University of California San Francisco (Site 203-001), San Francisco, California
  - Stanford University Hospital & Clinics (Site 203-003), Stanford, California
  - Lundquist Institute for Biomedical Innovation (Site 066-002), Torrance, California
  - Rocky Mountain Regional VA Medical Center (Site 074-010), Aurora, Colorado
  - University of Colorado Hospital (Site 204-001), Aurora, Colorado
  - Public Health Institute at Denver Health (Site 017-004), Denver, Colorado
  - Yale University (Site 025-001), New Haven, Connecticut
  - MedStar Health Research Institute/MedStar Washington Hospital Center (Site 009-021), Washington D.C., District of Columbia
  - Washington DC VA Medical Center (Site 009-004), Washington D.C., District of Columbia
  - University of Florida - Gainesville (Site 201-004), Gainesville, Florida
  - Miami VA Healthcare System (Site 074-003), Miami, Florida
  - Orlando VA Medical Center (Site 074-032), Orlando, Florida
  - Tampa General Hospital (032-001), Tampa, Florida
  - John H. Stroger, Jr. Hospital of Cook County (Site 080-046), Chicago, Illinois
  - University of Illinois at Chicago (Site 008-012), Chicago, Illinois
  - Carle Foundation Hospital (Site 080-049), Urbana, Illinois
  - Lutheran Medical Group (Site 301-010), Fort Wayne, Indiana
  - The University of Kansas Hospital (Site 080-044), Kansas City, Kansas
  - University of Kentucky (Site 210-004), Lexington, Kentucky
  - NIH Clinical Center (Site 080-043), Bethesda, Maryland
  - Massachusetts General Hospital (202-002), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Site 202-001), Boston, Massachusetts
  - Baystate Medical Center (Site 201-001), Springfield, Massachusetts
  - UMass Chan Medical School (Site 080-007), Worcester, Massachusetts
  - VA Ann Arbor Healthcare System (Site 074-028), Ann Arbor, Michigan
  - Henry Ford Health System (Site 014-001), Detroit, Michigan
  - Sinai-Grace Hospital (Site 205-005), Detroit, Michigan
  - Hennepin Healthcare Research Institute (Site 027-001), Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center (Site 112-001), Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic (Site 054-001), Rochester, Minnesota
  - University of Mississippi Medical Center (Site 202-005), Jackson, Mississippi
  - Washington University School of Medicine (Site 003-001), St Louis, Missouri
  - University of Nebraska Medical Center (Site 080-045), Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center (301-024), Lebanon, New Hampshire
  - Cooper University Hospital (Site 019-001), Camden, New Jersey
  - Hackensack Meridian Health (Site 301-030), Hackensack, New Jersey
  - New Jersey Medical School Clinical Research Center (028-001), Newark, New Jersey
  - University of New Mexico Hospital (Site 213-008), Albuquerque, New Mexico
  - CHRISTUS - St. Vincent (Site 080-051), Santa Fe, New Mexico
  - NYU Brooklyn (301-033), Brooklyn, New York
  - New York Presbyterian Queens (003-005), Flushing, New York
  - Mount Sinai Queens (Site 081-105), Long Island City, New York
  - NYU Long Island (301-034), Mineola, New York
  - New York University Tisch Hospital (Site 301-013), New York, New York
  - Mount Sinai Medical Center (Site 301-012), New York, New York
  - NYC Health + Hospital Harlem (Site 003-003), New York, New York
  - Weill Cornell Clinical Research Unit (065-001), New York, New York
  - St. Lawrence Health System (Site 301-029), Potsdam, New York
  - Lincoln Medical Center (Site 003-016), The Bronx, New York
  - Montefiore Medical Center - Moses Hospital (Site 206-001), The Bronx, New York
  - Montefiore Medical Center - Weiler campus (Site 206-003), The Bronx, New York
  - James J. Peters VAMC (Site 023-003), The Bronx, New York
  - Duke University Hospital (Site 301-006), Durham, North Carolina
  - Wake Forest Baptist Health (Site 210-001), Winston-Salem, North Carolina
  - University of Cincinnati Medical Center (Site 207-003), Cincinnati, Ohio
  - Cleveland Clinic Foundation (Site 207-001), Cleveland, Ohio
  - Ohio State University Wexner Medical Center (Site 207-004), Columbus, Ohio
  - Portland VA Health Care System (074-024), Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center (Site 209-002), Hershey, Pennsylvania
  - Rhode Island Hospital (Site 080-036), Providence, Rhode Island
  - The Miriam Hospital (Site 080-039), Providence, Rhode Island
  - Kent County Memorial Hospital (080-048), Warwick, Rhode Island
  - Ralph H. Johnson VA Medical Center (Site 074-015), Charleston, South Carolina
  - Medical University of South Carolina (Site 210-002), Charleston, South Carolina
  - Monument Health Rapid City Hospital (Site 213-005), Rapid City, South Dakota
  - Vanderbilt University Medical Center (Site 212-001), Nashville, Tennessee
  - Hendrick Medical Center (Site 080-014), Abilene, Texas
  - CHRISTUS Spohn Shoreline Hospital (Site 080-001), Corpus Christi, Texas
  - Baylor, Scott and White Health (301-003), Dallas, Texas
  - Parkland Health and Hospital Systems (Site 084-002), Dallas, Texas
  - UT Southwestern Medical Center (Site 084-001), Dallas, Texas
  - Houston Methodist Hospital (Site 301-028), Houston, Texas
  - MEDVAMC (Site 074-006), Houston, Texas
  - University of Texas Health Science Center (Site 203-006), Houston, Texas
  - CHRISTUS Good Shepherd Medical Center (Site 080-031), Longview, Texas
  - UT Health San Antonio (Site 009-022), San Antonio, Texas
  - Intermountain Medical Center (Site 211-001), Murray, Utah
  - University of Utah Health (Site 211-002), Salt Lake City, Utah
  - University of Virginia Health System, University Hospital (Site 210-003), Charlottesville, Virginia
  - Salem VA Medical Center (Site 074-014), Salem, Virginia
  - Harborview Medical Center (208-001), Seattle, Washington
  - Providence (Sacred Heart) (Site 213-004), Spokane, Washington
  - West Virginia University Medicine (301-023), Morgantown, West Virginia
  - William S. Middleton Memorial Veterans Hospital (074-030), Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital (052-001), Milwaukee, Wisconsin
- Argentina (7):
  - Instituto Medico Platense (Site 611-025), La Plata, Buenos Aires
  - Sanatorio Allende (Site 611-030), Córdoba, Córdoba Province
  - Clínica Central S.A. (611-028), Villa Regina, Río Negro Province
  - Sanatorio Británico S.A. (611-027), Rosario, Santa Fe Province
  - CEMIC (Site 611-021), Buenos Aires
  - Hospital Rawson (Site 611-012), Córdoba
  - Sanatorio Medico de Diagnostico y Tratamiento (611-029), Santa Fe
- Australia (5):
  - South Western Sydney Local Health District, Liverpool (Site 612-063), Liverpool, New South Wales
  - St. Vincent's Hospital (Site 612-002), Sydney, New South Wales
  - Westmead Hospital (Site 612-058), Westmead, New South Wales
  - Austin Health (612-020), Heidelberg, Victoria
  - The Alfred Hospital (Site 612-017), Melbourne, Victoria
- Brazil (12):
  - Fundação Universidade Caxias do Sul Hospital Geral (649-218), Caxias do Sul, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre (649-101), Porto Alegre, Rio Grande do Sul
  - Sociedade Literária e Caritativa Santo Agostinho - Hospital São José (Site 649-204), Criciúma, Santa Catarina
  - Hospital Nereu Ramos (Site 649-210), Florianópolis, Santa Catarina
  - Unimed Joinville Cooperativa de Trabalho Médico (Site 649-202), Joinville, Santa Catarina
  - Associação Beneficente Hospital Universitário - Universidade de Marília (Site 649-212), Marília, São Paulo
  - Instituto de Infectologia Emílio Ribas - IIER (Site 649-001), São Paulo, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência de São Paulo (Site 649-201, São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz (649-215), São Paulo, São Paulo
  - Associação Beneficente Síria - HCor (Site 649-203), São Paulo, São Paulo
  - Hospital SEPACO (649-207), São Paulo, São Paulo
  - Sociedade Beneficente de Senhoras Hospital Sirio-Libanês (Site 649-217), São Paulo, São Paulo
- Denmark (10):
  - Aarhus Universitetshospital, Skejby (625-002), Aarhus, N
  - Aalborg Hospital (Site 625-005), Aalborg
  - Rigshospitalet, CHIP (Site 625-006), Copenhagen
  - Bispebjerg Hospital (Site 625-013), Copenhagen
  - Herlev/Gentofte Hospital (Site 625-012), Hellerup
  - Nordsjaellands Hospital, Hillerod (Site 625-009), Hillerød
  - Hvidovre University Hospital, Department of Infections Diseases (Site 625-001), Hvidovre
  - Kolding Sygehus, Medicinsk Afdeling (Site 625-011), Kolding
  - Odense University Hospital (Site 625-004), Odense
  - Zealand University Hospital Roskilde (Site 625-010), Roskilde
- AIDS and Clinical Immunology Research Center (Site 627-201), Tbilisi, Georgia
- Germany (3):
  - Universitätsklinikum Bonn, Medizinische Klinik I, Immunologische Ambulanz (622-010), Bonn
  - Klinik I für Innere Medizin der Universität zu Köln (Site 622-008), Cologne
  - Johann Wolfgang Goethe Univ. Hosp., Infektionsambulanz CRS (622-001), Frankfurt
- Greece (5):
  - Dept of Critical Care and Pulmonary Medicine, Evangelismos General Hospital (635-020), Athens, Attica
  - 1st Respiratory Medicine Dept, Athens University Medical School (635-015), Athens, Attica
  - 3rd Dept of Medicine, Medical School (635-022), Athens, Attica
  - Attikon University General Hospital (Site 635-009), Athens, Attica
  - Democritus University of Thrace (635-021), Alexandroupoli, Evros
- Japan (3):
  - Fujita Health University Hospital (Site 612-105), Toyoake, Aichi-ken
  - Center Hospital of the National Center for Global Health and Medicine (Site 612-101), Shinjuku-Ku, Tokyo
  - Rinku General Medical Center (Site 612-107), Osaka
- Mexico (3):
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Site 653-001), Mexico City, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias Ismael Cosió Villegas (Site 653-002), Mexico City, Mexico City
  - Hospital General Dr. Aurelio Valdivieso (Site 653-004), Oaxaca City, OA
- Institute of Human Virology-Nigeria (IHVN) (Site 612-601), Abuja, Federal Capital Territory, Nigeria
- Peru (2):
  - Hospital Nacional Hipolito Unanue (651-008), Lima
  - Hospital Nacional Sergio E. Bernales (651-007), Lima
- Wojewodzki Szpital Zakazny (Site 625-302), Warsaw, Poland
- VA Caribbean Health Care (074-033), San Juan, PR, Puerto Rico
- Tan Tock Seng Hospital (Site 612-201), Singapore, Singapore
- South Africa (3):
  - Durban International Clinical Research Site (WWH) (652-005), Durban, KwaZulu-Natal
  - Greys Hospital (080-202), Pietermaritzburg, KwaZulu-Natal
  - University of Cape Town (UCT) Lung Institute (Site 080-201), Cape Town, Western Cape
- South Korea (4):
  - Seoul National University Bundang Hospital (Site 612-904), Seongnam-si, Gyeonggi-do
  - Seoul St. Mary's Hospital (Site 612-903), Seocho, Seoul
  - Asan Medical Center (612-901), Seoul
  - Chung-Ang University Hospital (Site 612-902), Seoul
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol (626-003), Badalona, Barcelona
  - Hospital del Mar (626-025), Barcelona
  - Hospital Universitari Vall d'Hebron (Site 626-033), Barcelona
  - Hospital Clinic de Barcelona (626-004), Barcelona
  - Hospital General Universitario Gregorio Marañón (Site 626-001), Madrid
  - Hospital Clínico San Carlos (Site 626-017), Madrid
  - Hospital Universitario La Paz (Site 626-012), Madrid
- University Hospital Zurich (Site 621-201), Zurich, Switzerland
- Thailand (2):
  - Chulalongkorn University and The HIV-NAT (Site 613-001), Bangkok
  - Khon Kaen University, Srinagarind Hospital (Site 613-003), Khon Kaen
- Uganda (5):
  - MRC/UVRI & LSHTM Uganda Research Unit (634-601), Entebbe
  - Gulu Regional Referral Hospital (634-603), Gulu
  - St. Francis Hospital, Nsambya (Site 634-607), Kampala
  - Lira Regional Referral Hospital (634-605), Lira
  - Masaka Regional Referral Hospital (634-606), Masaka
- Ukraine (3):
  - Central City Clinical Hospital of Ivano-Frankivsk City Council (Site 627-302), Ivano-Frankivsk
  - Treatment and Diagnostic Center ADONIS Plus (627-304), Kyiv
  - Hospital #1 of Zhytomyr City Council (627-303), Zhytomyr
- United Kingdom (3):
  - Royal Free Hospital (634-006), London
  - Guy's & St. Thomas' NHS Foundation Trust (Site 634-011), London
  - Royal Victoria Infirmary (Site 634-007), Newcastle upon Tyne
- Parirenyatwa General Hospital (Site 634-901), Harare, Zimbabwe